CLINICAL TRIAL: NCT01896089
Title: Prospective, Multicenter, Observational Registry Study to Determine if Enrollment in a Regional Kidney Paired Donor Exchange Program Improves the Overall Rate of Kidney Transplantation in Sensitized Patients, and Sensitized Patients Undergoing Desensitization Treatments.
Brief Title: Regional Kidney Paired Donor Exchange in Sensitized Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BiologicTx, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: KPD6172013
Record Dates: First submitted 2013-06-28; First posted 2013-07-11 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: The Rate of Kidney Transplants in Sensitized Patients.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a prospective, multi-center, observational study to determine if a combination of desensitization and enrollment in a regional kidney paired donor (KPD) exchange program improves the overall rate of kidney transplantation in sensitized patients.

ELIGIBILITY:
Inclusion Criteria:

* A. Potential Recipients must meet the following inclusion criteria:

  1. Willing and able to sign an informed consent form
  2. Must be at least 18 years old
  3. Meet all recipient selection criteria of the transplant center
  4. Listed on the deceased donor kidney waiting list for renal transplant at a participating center
  5. Potential recipients must:

Group 1: have one or more medically suitable donors who are ABO incompatible or HLA incompatible (defined as positive serologic cross-match); or

Group 2: have a medically suitable donor that is otherwise deemed incompatible due to age, size, or other mismatch by their respective transplant center; or

Group 3: be listed on the deceased donor waiting list for ≥ one year without an identifiable living donor and have a PRA% ≥ 60%

B. Potential Living Donors must meet the following inclusion criteria:

1. Must provide informed consent in accordance with the process outlined in the Informed Consent Requirements Section of the KPD Program Manual of Operations
2. Must be at least 18 years old
3. Meet all living donor selection criteria of the transplant center
4. Meet the evaluation requirements set forth in the Living Donor Evaluation Section of the KPD Program Operational Guidelines

Exclusion Criteria:

* C. Recipients

  1. Do not meet selection criteria of the transplant center
  2. Eligible compatible donor at the time of enrollment
  3. Inactive (not eligible to receive a kidney) on the deceased donor waitlist
  4. Pregnant or breast feeding

D. Donors

1. Unwilling or unable to provide informed consent
2. Have identified barriers to donation as set forth in the Living Donor Evaluation Section of the KPD Program Manual of Operations (Appendix A)
3. Must not be currently listed as a potential living donor for any other recipient registered in the KPD system
4. Pregnant or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 250 renal transplant candidates at 6 transplantation centers in the United States (northwest) will participate.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The rate of kidney transplant in sensitized patients following desensitization and enrollment in a regional kidney paired donor exchange program | 24 months
  The rate of kidney transplant in sensitized patients following desensitization and enrollment in a regional kidney paired donor exchange program will be summarized.

SECONDARY OUTCOMES:
Overall number of kidney transplants per center/region | 24 months
  To determine the overall number of kidney transplants per center/region.

OTHER OUTCOMES:
The overall number of KPD matches in the region | 24 months
Donor types (direct, paired exchange, altruistic) | 24 months
The overall number of KPD exchange recipients transplanted in the region | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Florence, MD, Principal Investigator — Swedish Medical Center; Andrew Weiss, MD, Principal Investigator — Virginia Mason Medical Center; Douglas Norman, MD, Principal Investigator — Oregon Health and Science University; Richard Carson, MD, Principal Investigator — Sacred Heart Medical Center (Spokane)
Locations (2):
- United States (2):
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington